CLINICAL TRIAL: NCT07138521
Title: Optimizing Linezolid Dosing in Patients With Advanced Renal Impairment: a Therapeutic Drug Monitoring-based Evaluation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Linezolid TDM
Record Dates: First submitted 2025-08-07; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Kidney Disease
Keywords: Linezolid; Therapeutic dose monitoring
MeSH Terms: conditions — Kidney Diseases | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Linezolid level within therapeutic range
  Interventions: Drug: Linezolid (IV and PO)
- Group 2 (Experimental): Above the therapeutic range and within the toxicity range
  Interventions: Drug: Linezolid (IV and PO)
- Group 3 (Experimental): Above the therapeutic range and within the toxicity range
  Interventions: Drug: Linezolid (IV and PO)

INTERVENTIONS:
Drug: Linezolid (IV and PO) — No dose change and continued linezolid 600 mg every 12 hours.
  Other Names: 600-twice
  Arms: Group 1
Drug: Linezolid (IV and PO) — Intervention and adjustment of the linezolid dose from 600 mg every 12 hours to 300 mg every 12 hours.
  Other Names: 300-twice
  Arms: Group 2
Drug: Linezolid (IV and PO) — Intervention and adjustment of the linezolid dose from 600 mg every 12 hours to 600 mg every 24 hours.
  Other Names: 600-once
  Arms: Group 3

SUMMARY:
The goal of this clinical trial is to adjust the Linezolid dose according to its blood level in adults with kidney diseases. It will also learn about the safety of linezolid. The main questions it aims to answer are:

* How often does linezolid require level monitoring?
* How often does linezolid require dose adjustment?
* What medical benefits do participants have when linezolid level monitoring is applied? Researchers will compare two dose reduction regimens when they have evidence of overexposure to determine which regimen is more effective in preventing thrombocytopenia (Platelet drop).

Participants will:

* Withdrew linezolid level every 2 to 4 days of the antibiotic course.
* Visit the clinic twice for checkups and tests.

DETAILED DESCRIPTION:
Linezolid is a crucial antibiotic prescribed for the treatment of various infectious diseases such as pneumonia, skin infections, and catheter-related bloodstream infections. Linezolid covers gram-positive bacteria, including Methicillin-resistant Staphylococcus Auris (MRSA) and Vancomycin-resistant Staphylococcus Auris (VRSA).

Recently, Linezolid usage has become favorable for chronic kidney disease (CKD) patients to preserve the remaining residual renal function by avoiding nephrotoxic antibiotics such as vancomycin and aminoglycosides. However, linezolid-induced thrombocytopenia hinders linezolid use in the CKD population due to accumulation and overexposure. Recent literature suggested implementing a therapeutic drug monitoring (TDM) approach to modify the dose regimen and minimize linezolid toxicity.

The obstacle faced was the lack of clear TDM-based linezolid modification guidelines for CKD patients. To overcome this issue, we conducted a pilot study involving 15 patients (7 ESRD, 5 CKD, and 3 AKI on top of CKD). Patients with evidence of toxic levels (8 patients) underwent dose adjustment from 600mg every 12 hours to 300mg every 12 hours.

Dose reduction by 50% with no change in dose interval resulted in a decrease in supratherapeutic trough levels. However, these levels, while lower, did not consistently reach the predefined target therapeutic range (2-8 mg/dl).

The recent approach we are investigating now is to both lower the dose and elongate the interval.

The aim of the work is to optimize renal dosing adjustment with patients having linezolid by investigating whether once-daily dosing administration of linezolid provides better trough-range targeting over twice-daily targeting.

Research Steps

1. Patients were interviewed and selected according to the study's selection criteria.
2. Blood tests were taken before the start of the study to assess their condition and record their medical history before starting linezolid treatment.
3. Participants were divided into three groups based on linezolid drug concentrations compared to the pre-defined target therapeutic range, as determined by the pharmacotherapy monitoring guidelines:

   I. Group 1: Within the therapeutic range: No intervention and continued linezolid 600 mg every 12 hours.

   II. Group 2: Above the therapeutic range and within the toxicity range: Intervention and adjustment of the linezolid dose from 600 mg every 12 hours to 300 mg every 12 hours.

   III. Group 3: Above the therapeutic range and within the toxicity range: Intervention and adjustment of the linezolid dose from 600 mg every 12 hours to 600 mg every 24 hours.
4. Patient follow-up was conducted at the end of the study and comparisons were made between the different groups.

ELIGIBILITY:
Inclusion Criteria:

* Advanced renal impairment, Hemodialysis patients

Exclusion Criteria:

* Pregnancy, Lactating females, Advanced Liver impairment, Cases using antidepressants or antipsychotics, Cases suffering from Hematological blood diseases, and/or chronic Immune thrombocytopenia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Therapeutic range trough targeting | From enrollment to the end of antibiotic treatment duration (typically 10 to 14 days)
  Linezolid Therapeutic Range Trough Targeting - The proportion of patients whose steady-state linezolid trough concentrations fall within the predefined therapeutic range (e.g., 2-8 mg/L) during treatment as a result of level monitoring and dose correction. This range is the established range for antimicrobial efficacy while minimizing the risk of toxicity, particularly hematological adverse effects. Concentrations will be measured using validated analytical method using HPLC device, and results will be compared to target thresholds to evaluate dosing adequacy.

SECONDARY OUTCOMES:
Incidence of New-Onset Thrombocytopenia | From enrollment to the end of antibiotic treatment duration (typically 10 to 14 days)
  Proportion of participants (Unit of Measure: % of participants) who develop new-onset thrombocytopenia during linezolid therapy, defined as a platelet count <150 × 10⁹/L or a ≥25% reduction from baseline, whichever is lower.
  Platelet counts (× 10⁹/L) will be monitored at baseline and predetermined intervals throughout therapy and obtained through routine laboratory testing.
Correlation Between Linezolid Trough Concentrations and Thrombocytopenia | From enrollment to the end of antibiotic treatment (typically 10-14 days).
  Correlation analysis of linezolid trough concentrations with thrombocytopenia occurrence: The measurement tools are plasma trough concentration of linezolid (mg/L, measured by validated HPLC) and platelet count (× 10⁹/L, measured by routine laboratory testing). The relationship will be assessed using correlation coefficient (r) calculations.

IPD SHARING:
Plan to Share IPD: Yes
Variables including: Age, Weight, Gender, Blood workups, such as Platelets count and Linezolid blood levels.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Start date: Once recruitment is completed and required data is collected. End date: Paper publishing date.
Access Criteria: Study supervisors and co-researchers will have access for data interpretation and analysis once collected.

REFERENCES:
- See also: Dose optimisation of linezolid in critically ill patients based on a population pharmacokinetic model: A two-centre prospective interventional study — https://pubmed.ncbi.nlm.nih.gov/37301313
- See also: Pharmacokinetics of Linezolid Dose Adjustment for Creatinine Clearance in Critically Ill Patients: A Multicenter, Prospective, Open-Label, Observational Study — https://pubmed.ncbi.nlm.nih.gov/34040351
- See also: Dosage Strategy of Linezolid According to the Trough Concentration Target and Renal Function in Chinese Critically Ill Patients — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9035989
- See also: Reappraisal of Linezolid Dosing in Renal Impairment To Improve Safety — https://pubmed.ncbi.nlm.nih.gov/31109977
- See also: Analysis of thrombocytopenic effects and population pharmacokinetics of linezolid: a dosage strategy according to the trough concentration target and renal function in adult patients — https://pubmed.ncbi.nlm.nih.gov/25108880